CLINICAL TRIAL: NCT00725868
Title: Blood Endothelium Biomarkers to Predict Major Adverse Cardiovascular Events After Percutaneous Coronary Intervention.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Assistance Publique Hopitaux De Marseille, Assistance Publique Hopitaux De Marseille
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2007-A00533-50; 2007-18
Record Dates: First submitted 2008-07-30; First posted 2008-07-31 (Estimated); Last update posted 2011-08-26 (Estimated); Status verified 2011-08

CONDITIONS: Atherosclerosis; Percutaneous Coronary Intervention; Cardiovascular Diseases
Keywords: Major adverse
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases | interventions — Angioplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): Data private hospitals, angioplasty, sampling of blood
  Interventions: Other: Data private hospitals, angioplasty, sampling of blood

INTERVENTIONS:
Other: Data private hospitals, angioplasty, sampling of blood — * Data private hospitals : Age, sex, index of body mass, factors of cardiovascular risk, medical surgical histories, treatment before and after the angioplasty, the renal insufficiency
  * coronary angioplasty
  * Sampling of blood : Before the angioplasty, 6 hours after the angioplasty and 24 hours after the angioplasty. A numeration of the proparents circulants (hématopoietics, PEC) and a numeration of CEC are made

SUMMARY:
In stent restenosis and myocardial infarction are have been linked the balance between injury and healing of the endothelium These processes can be measured respectively using the number of circulating endothelial cells and endothelial progenitor cells. We therefore aimed to evaluate the relationship between the balance of injury and healing of the endothelium at the time of PCI and major adverse cardiovascular events including death, myocardial infarction and target lesion revascularization at 6 and 12 months follow-up.

DETAILED DESCRIPTION:
Following percutaneous coronary intervention with bare metal stents, the rate of major adverse cardiovascular events including death, myocardial infarction and target lesion revascularization is high ranging between 20 and 25%.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years old
* Scheduled for PCI
* Clinical evidence of ischemic heart disease and/or abnormal functional study
* New coronary artery lesion >50%
* treatment with bare metal stent planned
* Informed consent explained, red, understood and signed by the patient

Exclusion Criteria:

* Pregnancy, birth or lactation period <6 months ago
* Women of childbearing age who do not intend to use accepted anticonceptive measures or who wish to get pregnant
* Left ventricular ejection fraction <30%
* Acute coronary syndrome (ST-elevation or not) in the past month
* Planned drug eluting stent implantation
* Lesion in arterial or venous bypass or anastomosis with coronary
* Severe renal insufficiency (creatinine clearance <30 mL/')
* Severe hepatic insufficiency
* Systemic inflammatory pathology of any kind
* Hematologic or other malignancy, prior radio- or chemotherapy
* Use of corticosteroïds or immune suppression therapy
* Contrast allergy
* Life expectancy <1 year
* Participation in other clinical study which has not ended yet

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2007-09; Primary Completion 2010-08 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
The main objective of this study is to estimate if the measure of CEC and PEC possesses a meaning forecast towards the arisen of complications post procedure. | 36 months

SECONDARY OUTCOMES:
To determine the relation between these endothelial biomarkers and the other usual parameters forecast complications post-angioplasty | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Franck PAGANELLI, MD, Principal Investigator — Assistance Publique des Hopitaux de Marseille
Locations (1):
- Service de Cardiologie- Hopital Nord, Marseille, France